CLINICAL TRIAL: NCT01557205
Title: Research and System Development on Functional 3D Optical Tomography for Skin Cell Imaging
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Professor, National Taiwan University
Other Study IDs: 201202019RIC
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Optical Coherence Tomography; Skin Cell Imaging
Keywords: optical coherence tomography; cell imaging

STUDY DESIGN:
Biospecimen Retention: None Retained — No biospecimen to be retained.
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will obtain human skin specimen (sized approximately 1 cm x 1 cm) for dermatological surgical patients in National Taiwan University Hospital, after informed consent was obtained. Human skin keratinocytes, fibroblasts, and melanocytes will be cultured from the human skin specimen. The three dimensional images of these cultured cells will be observed by a ultra-high resolution 3-dimensional optical coherence tomography.

DETAILED DESCRIPTION:
The investigators will obtain human skin specimen (sized approximately 1 cm x 1 cm) for dermatological surgical patients in National Taiwan University Hospital, after informed consent was obtained. Human skin keratinocytes, fibroblasts, and melanocytes will be cultured from the human skin specimen. The three dimensional images of these cultured cells will be observed by a ultra-high resolution 3-dimensional optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 to 100.
* People who received benign skin tumor removal in dermatological surgical unit. OR
* People who received skin grafts (full thickness or split thickness) for reconstruction of surgical wounds after removing malignant skin cancer.

Exclusion Criteria:

* Age less than 20 years old,
* Psychiatric patients,
* Pregnant women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aged between 20 to 100. People who received benign skin tumor removal in dermatological surgical unit. OR people who received skin grafts (full thickness or split thickness) for reconstruction of surgical wounds after removing malignant skin cancer.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)